CLINICAL TRIAL: NCT05586191
Title: Effects of Home Versus Hospital Based Action Observation Therapy on Balance, Mobility and Cognition in Diaplegic Cerebral Palsy
Brief Title: Home Versus Hospital Based Action Observation Therapy in Diaplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HADIA HADI REC 01335
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Diplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation therapy at home (Experimental): In action observation therapy, patient will not come to hospital for treatment. He will see a video at home in which therapist will perform different activities then patient will also perform the same movements.
  Interventions: Other: Action observation at home
- Action Observation therapy at hospital (Active Comparator): In action observation therapy, patient will come to hospital for treatment. He will see a video in which therapist will perform different activities then patient will also perform the same movements.
  Interventions: Other: Action Observation therapy at hospital

INTERVENTIONS:
Other: Action observation at home — Exercises included will contain four stages of exercises. Each stage will be followed for 2 weeks i.e. stage 1 for 1st and 2nd week, second stage for 3rd and 4th week, third stage for 5th and 6th week and fourth stage for 7th and 8th week of treatment. Each component of every stage will be played for 1 minute in front of participants, followed by 1 minute rest and then these exercises will be performed for 5 minutes.
  All participants will perform AOT 3 times/week for up to 8 weeks along with functional training for the rest of the weeks. Functional training will include stretching and isometric exercises (stretching of hamstring and calf muscle while quads isometric). Assessment will be done by using the tools at baseline and after 8 weeks of intervention. A final reading will be taken after 12 weeks to check the maintenance of training effects.
  Other Names: stretching exercises of lower limb
  Arms: Action Observation therapy at home
Other: Action Observation therapy at hospital — Exercises included will contain four stages of exercises. Each stage will be followed for 2 weeks i.e. stage 1 for 1st and 2nd week, second stage for 3rd and 4th week, third stage for 5th and 6th week and fourth stage for 7th and 8th week of treatment. Each component of every stage will be played for 1 minute in front of participants, followed by 1 minute rest and then these exercises will be performed for 5 minutes.
  All participants will perform AOT 3 times/week for up to 8 weeks along with functional training for the rest of the weeks. Functional training will include stretching and isometric exercises (stretching of hamstring and calf muscle while quads isometric). Assessment will be done by using the tools at baseline and after 8 weeks of intervention. A final reading will be taken after 12 weeks to check the maintenance of training effects.
  Other Names: stretching exercises of lower limb
  Arms: Action Observation therapy at hospital

SUMMARY:
Effects of Home Versus Hospital Based Action Observation Therapy on Balance, Mobility and Cognition in Diaplegic Cerebral Palsy. It will be a RCT we want to identify the effects of action observation therapy on patients coming to the hospital as compared to the patients at home. We will also identify the retaining effects of AOT. Our sample size will be 40 diplegic patients having no cognitive issues and able to walk with assistive device. We will exclude the patient who will suffer with severe comorbidities and visual impairment. We will randomly assign the patients into two groups A and B.A will receive Action observation therapy three times a day along with stretching exercises .while group B we perform AOT and stretching exercises at home with same frequency.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category will be recruited into the study.

  * Diagnosed Diaplegic CP Children between the age of 5 to 11 years.
  * Without visual impairment and visual field defects.
  * Able to follow the researcher's instruction.
  * GMFCS (gross motor function classification system) level I-III.

Exclusion Criteria:

* Participants failing to fall in this category will be excluded of the study.

  * Children with a Modified Ashworth scale (MAS) of 3 or more
  * Unable to walk
  * Children with severe co-morbidities. (2)

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function measure (GMFM) | 12 weeks
  Changes from baseline,It is the valid and standard observational instrument to measure change in gross motor function in CP children. It consists of 66 items with 5 dimensions. These dimensions are the major motor functions i.e. supine/rolling, sitting, crawling/kneeling, standing and walking/running/jumping. Each task is rated according to the scoring guidelines i.e. higher score indicated better gross motor function. Each GMFM item is graded on 4-point scale i.e. 0 for unable to initiate the task, 1 for able to initiate the task, 2 for able to perform the task partially and 3 for able to perform the task completely. At the end these score summed up into total score.(21)
Pediatric Balance Scale (PBS) | 12 weeks
  Changes from baseline, It is a modified form of Berg Balance Scale (BSS) which was developed for balance measurement in CP child. It can be performed without specialized equipment and can be easily administered. It including 14 items with 5-level grading to assess the functional activities that child must safely and independently form at home, community, activities including sitting balance, sit to stand/stand to sit, transfer, stepping, reaching forward, reaching to floor, turning and stepping on and off at elevated surface. Each activity is rated according to scale from 0 to 4 i.e. 0 for unable to perform and 4 for able to perform without difficulty.
Timed 10 meter walk test | 12 weeks
  Changes from Baseline ,It was used to measure the gait ability and speed. The acceleration area 2.5m and deceleration area 2.5m were marked on the ground as start and end point for the test. Participants were asked to walk for 15 minutes on comfortable flat floor at a comfortable speed and then record the walking speed through stopwatch over 10 m between these point. The mean value of the three trials was used and expressed as m/s
Mini-mental state pediatric examination (MMSPE) | 12 weeks
  Changes from Baseline, it is a cognitive screening task and scoring system for 3 to 14 years old child. It represented 11 questions involving five basic cognitive abilities i.e. attention-concentration, orientation, registration, recall and language and constructive ability.(22) The possible score range is from 0 to 37, from which 17 or lower score indicating as moderate to severe cognitive impairment of children.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Bashir, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Irfan General Hospital Peshawar, Peshawar, Khyberpakhtunkhuwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeong YA, Lee BH. Effect of Action Observation Training on Spasticity, Gross Motor Function, and Balance in Children with Diplegia Cerebral Palsy. Children (Basel). 2020 Jun 18;7(6):64. doi: 10.3390/children7060064. PMID 32570855
- [Background] Numanoglu A, Gunel MK. Intraobserver reliability of modified Ashworth scale and modified Tardieu scale in the assessment of spasticity in children with cerebral palsy. Acta Orthop Traumatol Turc. 2012;46(3):196-200. doi: 10.3944/aott.2012.2697. PMID 22659636
- [Background] Kim Y, Lee BH. Clinical Usefulness of Child-centered Task-oriented Training on Balance Ability in Cerebral Palsy. J Phys Ther Sci. 2013 Aug;25(8):947-51. doi: 10.1589/jpts.25.947. Epub 2013 Sep 20. PMID 24259891
- [Background] Reid SM, Carlin JB, Reddihough DS. Distribution of motor types in cerebral palsy: how do registry data compare? Dev Med Child Neurol. 2011 Mar;53(3):233-8. doi: 10.1111/j.1469-8749.2010.03844.x. Epub 2010 Dec 17. PMID 21166669
- [Background] Joung HJ, Park J, Ahn J, Park MS, Lee Y. Effects of creative dance-based exercise on gait performance in adolescents with cerebral palsy. J Exerc Rehabil. 2020 Aug 25;16(4):332-343. doi: 10.12965/jer.2040384.192. eCollection 2020 Aug. PMID 32913838
- [Background] Oskoui M, Coutinho F, Dykeman J, Jette N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080. Epub 2013 Jan 24. PMID 23346889
- [Background] Park EC, Hwangbo G. The effects of action observation gait training on the static balance and walking ability of stroke patients. J Phys Ther Sci. 2015 Feb;27(2):341-4. doi: 10.1589/jpts.27.341. Epub 2015 Feb 17. PMID 25729163
- [Background] Ryan D, Fullen B, Rio E, Segurado R, Stokes D, O'Sullivan C. Effect of Action Observation Therapy in the Rehabilitation of Neurologic and Musculoskeletal Conditions: A Systematic Review. Arch Rehabil Res Clin Transl. 2021 Jan 27;3(1):100106. doi: 10.1016/j.arrct.2021.100106. eCollection 2021 Mar. PMID 33778479